CLINICAL TRIAL: NCT04137965
Title: Testicular Function After Testicular Torsion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Frederik Møller Jacobsen, Principal Investigator, Herlev and Gentofte Hospital
Other Study IDs: Torsion study
Record Dates: First submitted 2019-10-18; First posted 2019-10-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Testicular Torsion; Spermatic Cord Torsion
Keywords: Fertility; Testicular Torsion; Testicular function
MeSH Terms: conditions — Spermatic Cord Torsion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Testicular torsion group: Men having undergone surgery for testicular torsion between 01.01.2003 and 12.31.2012
- Control group: Men without knowledge of their fertility status and who have never had their semen analyzed

SUMMARY:
The purpose of this study is to evaluate testicular function measured as testosterone level and semen quality.

DETAILED DESCRIPTION:
Men having undergone surgery for testicular torsion between 01.01.2003 - 12.31.2012 will receive a invitation to participate in this study. It is expected that 110 patients can be identified and about 65% of them will participate. These men will undergo a andrological evaluation, deliver a semen sample, have a blood sample taken and undergo a testicular ultrasound.

Control group:

Men attending the fertility counseling at Herlev hospital will be offered participation in this study. The fertility counseling demands that men who contact the clinic have never had their sperm analyzed, have not tried to get pregnant with their partner for more than a year and that they have no prior knowledge of their fertility.

Primary endpoint:

* Semen quality measured as sperm concentration
* Total testosterone level

Secondary endpoint:

Semen parameters

* Semen volume (ml)
* Sperm concentration (x 106/ml)
* Sperm motility (%) (både klasse AB og ABC)
* sperm morphology
* IgA-bound spermatozoa (%)
* IgG-bound spermatozoa (%)

Hormones

* FSH
* LH
* PRL
* Testosterone
* Estradiol
* Inhibin B
* Insulin-like peptide 3
* SHBG

Data points:

* Paternity
* Time to pregnancy
* Partner (yes/no)
* Any fertility treatment?
* Pain? (VAS score)
* Symptoms of testesterone deficiency symptoms
* Andrological evaluation
* Testicular ultrasound
* Testicular torsion events in the family
* Date of surgery
* Date of follow up meeting
* Surgery details

ELIGIBILITY:
Inclusion Criteria:

* Men with a verified testicular torsion operated at Herlev and Gentofte hospital between 01.01.2003 and 12.31.2012

Exclusion Criteria:

* Retentio testis
* Varicocele
* Previous treatment with chemo- or radiation therapy
* Genetic disposition for infertility
* Anejculation
* Retrograde ejaculation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with a verified testicular torsion operated at Herlev and Gentofte hospital between 01.01.2003 and 12.31.2012. This ensures atleast 5 years of follow up.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Sperm concentration | 8-17 years after surgical intervention
  Amount of motile sperm cells (* 10^6)
Testosterone level | 8-17 years after surgical intervention
  ng/ml

SECONDARY OUTCOMES:
Semen parameters as an indicator of overall testicular exocrine function | 8-17 years after surgical intervention
  Compared with results from control group
Hormone level as an indicator of testicular endocrine function | 8-17 years after surgical intervention
  Follicle stimulating hormone, luteinizing hormone, prolactin, testosterone, estradiol, inhibin B, sex hormone-binding globulin, albumin
MAR test result correlated to the type of surgery | 8-17 years after surgical intervention
  MAR test of sperm cells
Difference in sperm morphology and motility correlated to the type of surgery and compared to control group | 8-17 years after surgical intervention
  Morphology and motility (%)
Paternity as a measure of fertility | 8-17 years after surgical intervention
  Number of kids if any.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Sønksen, Professor, Study Director — Herlev and Gentofte Hospital
Locations (1):
- Department of Growth and Reproduction, Copenhagen, Denmark